CLINICAL TRIAL: NCT07127575
Title: A Scalable Intervention for Stress Management Practices
Brief Title: Scalable Intervention for Stress Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Livotion, LLC (Industry)
Collaborators: Purdue University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-935; 1R41AT012854-01 (NIH)
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Stress; Diaphragmatic Breathing
Keywords: resistance breathing; stress management

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three conditions. 20 will be in the no pen condition, 20 will be in the original AIRpen condition, and 20 will be in the smart AIRpen condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Base AIRpen (Experimental): In this arm, participants will utilize an AIRpen after completing an arithmetic based stress test during a decompression period. Participants will engage in diaphragmatic breathing and other stress reducing behaviors like fidgeting or clicking using the AIRpen while physiological data is measured with an ear sensor and audio recordings.
  Interventions: Device: Resistance Breathing Device
- Smart AIRpen (Experimental): In this arm, participants will utilize a SMART AIRpen after completing an arithmetic based stress test during a decompression period. Participants will engage in diaphragmatic breathing and other stress reducing behaviors like fidgeting or clicking using the Smart AIRpen while physiological data is measured with an ear sensor and audio recordings.
  Interventions: Device: Electronic Resistance Breathing Device
- No AIRpen (No Intervention): In this arm, participants will be asked to sit quietly following an arithmetic based stress test during a decompression period. Physiological data will be measured with an ear sensor and audio recordings.

INTERVENTIONS:
Device: Resistance Breathing Device — The AIRpen is a multifunctional stress management tool that helps users engage in diaphragmatic breathing at differing resistance levels, as well as other common stress relieving behaviors such as fidgeting
  Arms: Base AIRpen
Device: Electronic Resistance Breathing Device — The Smart AIRpen functions just as the original AIRpen device and has been augmented with sensors to measure use patterns to determine whether the AIRpen is being used for fidgeting or breathing.
  Arms: Smart AIRpen

SUMMARY:
The purpose of this research is to measure the acceptance of a resistance breathing intervention and to assess whether it produces physiological and subjective effects in a laboratory setting.

DETAILED DESCRIPTION:
College students experience a wide range of stressors during their studies, with many students experiencing levels of stress that can be clinically significant, such as anxiety or depression. Counseling centers on college campuses have seen a rise in students seeking mental health support or stress relief, but there exists a discrepancy in the level of need versus the support that can be provided. Stress management interventions, such as self-care mobile applications and devices, have risen in popularity given their relative accessibility and implementation of stress relieving interventions such as regulated breathing. Regulated breathing has been shown to be a reliable and effective form of stress relief, however its implementation within various eHealth interventions and related devices can come into conflict when used in educational settings. Mobile apps and biofeedback devices (e.g., chest straps, inhalers), can be contextually inappropriate, cumbersome, and potentially stigmatizing for students. To overcome these barriers, the PI developed the AIRpen, a simple, affordable, multi-functional stress management device that is designed to fit into the fabric of students' lives to potentially optimize the delivery, practice, and fidelity of diaphragmatic breathing (DB) interventions in real- world settings. With anecdotal and empirical evidence supporting the device as feasible and acceptable in real-world academic settings, this study will build upon prior work and measure the acceptance of the intervention and assess whether using the original and a "smart" version of the device as a stress relieving tool produces physiological and subjective effects in a laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be currently enrolled in a college or university
* Be able to read, speak, and comprehend English
* Be able and willing to complete a 60-minute study involving heart rate monitoring, survey completion, training, a stress test, and device utilization

Exclusion Criteria:

-Individuals diagnosed with anxiety or stress and require professional support to cope with these clinical levels of stress or anxiety should not enroll in the study in place of professional assistance.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Device Acceptability as Measured by the Acceptability of Intervention Measure (AIM) | From enrollment to end of 1 hour study period.
  The AIM measure is designed to assess the acceptability of a intervention, and has been adapted in relation to the AIRpen. Participants rate statements related to their usage and experience of the AIRpen and AIRpen website, with ratings ranging from "Completely Disagree" (1), to "Completely Agree" (5). Higher scores indicate higher acceptability of the intervention.
Device Usability as Measured by a Modified Version of the System Usability Scale (SUS) | From enrollment until completion of 1 hour study period.
  The System Usability Scale is a 10-item measure that address the usability and learnability of a system. The SUS has been modified to reflect the AIRpen intervention. Statements are ranked on a Likert scale for 1-5, with 1 indicating "Strongly Disagree" and 5 indicating "Strongly Agree". Raw scores are converted into a final score that ranges from 0-100, with a larger score indicating greater usability.

SECONDARY OUTCOMES:
Perceived Stress as Measured by the Perceived Stress Scale (PSS_10) | From enrollment to the end of the 1 hour study period
  The Perceived Stress Scale is a measure used to assess perceptions of recent stress. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Physiological Stress as Assessed with Heart Rate Monitoring | From study enrollment to end of 1 hour study period

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No